CLINICAL TRIAL: NCT06011902
Title: A 6-month Follow-up Study of Patients With Severe Fever With Thrombocytopenia Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qin Ning, Director and Chair of Department of Infectious Diseases, Tongji Hospital
Other Study IDs: RESORT
Record Dates: First submitted 2023-08-08; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Severe Fever With Thrombocytopenia Syndrome
MeSH Terms: conditions — Severe Fever with Thrombocytopenia Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This is a multi-center, retrospective clinical study to analyze the clinical features, laboratory indicators, imaging changes, treatment options and long-term prognosis in patients with sever fever with thrombocytopenia syndrome. All hospitalized patients with sever fever with thrombocytopenia diagnosed between 2016 and 2022 were included from the electronic medical record system of 8 centers, and demographics, hospitalization information, clinical information, laboratory or imaging examinations, treatment options, and outcomes were collected.

ELIGIBILITY:
Inclusion Criteria:

* Age and gender are not limited;
* Hospitalized patients diagnosed with severe fever with thrombocytopenia syndrome have at least one of the following laboratory test results: serum severe fever with thrombocytopenia syndrome bunyavirus (SFTSV)-specific IgM antibody positive or IgG antibody level increased more than 4 times; or positive for SFTSV RNA; or positive for SFTSV nucleic acid detected by real-time fluorescent quantitative RT-PCR; or SFTSV isolated from case specimens.

Exclusion Criteria:

* Patients who were found to be positive for other tick-borne pathogens by PCR analysis of blood samples in the acute phase;
* It is difficult to conduct outpatient follow-up due to mental disorders, dementia, combined diseases such as osteoarthropathy, stroke, pulmonary embolism, etc. that lead to inability to move freely;
* No outpatient follow-up visit after discharge, and repeated confirmation by phone call still unable to get in touch;
* Due to living in other places, nursing homes, welfare homes, unable to participate in outpatient follow-up after making an appointment by phone;
* Currently participating in clinical trials of other drugs or medical devices;
* The researchers think it is not suitable for inclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients diagnosed with severe fever with thrombocytopenia syndrome from 8 centers in Hubei Province, China.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
The presense of clinical symptoms of patients at 3 months and 6 months after discharge | 3 months,6 months
  The number and severity of clinical symptoms of patients.

SECONDARY OUTCOMES:
Number of participants with different outcome of disease | 6 months
  Number of participants who experience these events:
  1. discharge with improvement
  2. death
  3. automatic discharge

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - NO.1 Peoples Hospital of Guangshui, Guangshui, Hubei
  - Huanggang Central Hospital, Huanggang, Hubei
  - People's Hospital Of Luotian County, Huanggang, Hubei
  - People's Hospital of Macheng city Affiliated Hospital of Hubei Univerciy of science and technology, Macheng, Hubei
  - Suizhou Central Hospital, Suizhou, Hubei
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xianning Central Hospital, Xianning, Hubei
  - Yichang Third Peoples Hospital, Yichang, Hubei